CLINICAL TRIAL: NCT02967783
Title: A Pragmatic Trial to Quantitatively and Qualitatively Assess Different Techniques for the ID Administration of Fractional Dose IPV in a Campaign Setting in The Gambia
Brief Title: A Campaign-based ID fIPV Administration Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Research Council Unit, The Gambia (Other)
Collaborators: World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: London School of Hygiene and Tropical Medicine (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SCC1495
Record Dates: First submitted 2016-09-19; First posted 2016-11-18 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Needles; Syringes

STUDY DESIGN:
Masking Description: six vaccination teams will be randomly assigned to administer the three different ID fIPV administration technique the campaign days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ID Needle and Syringe (Active Comparator): Fractional (0.1mL) dose of inactivated poliovirus vaccine (IPV) administered using a needle and syringe
  Interventions: Device: Needle and syringe
- ID Adaptor (Helm) (Experimental): Fractional (0.1mL) dose of inactivated poliovirus vaccine (IPV) administered using a needle and syringe with an ID adaptor
  Interventions: Device: ID adaptor
- ID Jet Injector (Tropis, Pharmajet) (Experimental): Fractional (0.1mL) dose of inactivated poliovirus vaccine (IPV) administered by needle and syringe with a disposable syringe jet injecto
  Interventions: Device: ID Jet Injector (Tropis, Pharmajet)

INTERVENTIONS:
Device: ID adaptor — ID adaptor fixed to the end of a standard ID needle and syringe to facilitate ID administration of the inactivated poliovirus vaccine
  Arms: ID Adaptor (Helm)
Device: ID Jet Injector (Tropis, Pharmajet) — ID disposable syringe (needle free) jet injector to facilitate ID administration of the inactivated poliovirus vaccine
  Arms: ID Jet Injector (Tropis, Pharmajet)
Device: Needle and syringe — Standard ID needle and syringe for ID administration of the inactivated poliovirus vaccine
  Arms: ID Needle and Syringe

SUMMARY:
The introduction of one dose of the inactivated poliovirus vaccine (IPV) into routine immunization schedules in OPV-only using countries as part of the Global Polio Eradication Initiative (GPEI) was planned for completion in 2016. However, due to recent developments in the global IPV supply landscape, the GPEI polio eradication program is facing a critical shortage of the vaccine which is forecast to continue until at least the end of 2017. The shortage means that some countries that have already introduced the vaccine, but which are considered to be relatively low risk (The Gambia included), will be left without adequate supplies and in other countries IPV introduction is being unavoidably delayed.

Exacerbating the shortage is the need to reserve IPV for future outbreak responses (OBR). The current OBR protocol recommends that, if a circulating vaccine-derived poliovirus type 2 (cVDPV2) outbreak occurs (after the recent global switch from trivalent to bivalent OPV), a large scale IPV campaign will be implemented to increase population immunity to the type 2 poliovirus in an large area surrounding the outbreak as high risk of extending transmission.

Due to above, dose-sparing through the administration of intra-dermal (ID) fractional (one fifth - 0.1mL) doses of IPV (fIPV) has become a very important focus and, for planning purposes, there is an urgent need to assess the practical and logistic challenges a country such as The Gambia would face in rapidly undertaking an ID fIPV campaign.

DETAILED DESCRIPTION:
Background information and rationale

Background information

Polio eradication requires the removal of all polioviruses from the human population, whether wild-type poliovirus (WPV) or those vaccine-derived polioviruses (VDPV) emanating from the oral poliovirus vaccine (OPV). The Polio Eradication & Endgame Strategic Plan 2013-2018 provides a framework for interruption of WPV transmission in remaining endemic foci and lays out plan for the new polio endgame. This will include the withdrawal of Sabin strains, starting with the type 2 strain, and the introduction of the inactivated poliovirus vaccine (IPV), for risk mitigation purposes.

The introduction of one dose of IPV into routine immunization schedules in OPV-only using countries was planned for completion in 2016. However, due to recent developments in the global IPV supply landscape, the polio eradication program is facing a critical shortage of the vaccine which is currently forecast to continue until at least the end of 2017. The shortage is not only preventing the universal introduction of one dose of IPV into some routine immunization schedule but may also mean that some countries who have already introduced the vaccine, but are considered to be relatively low risk, will be left without adequate supplies.

Exacerbating the shortage is the demand to reserve IPV for future outbreak responses (OBR). The current OBR protocol recommends that, in the event of a circulating vaccine-derived poliovirus type 2 (cVDPV2) outbreak after the switch, a large scale IPV response is implemented - a preventive campaign in the zone surrounding the outbreak (rather than the core area of the outbreak itself) to increase population immunity to the type 2 poliovirus in an area at high risk of driving further transmission considering the ongoing VDPV2 outbreak nearby.

In light of the number of individuals to be vaccinated under such circumstances, dose-sparing through the administration of intradermal (ID) fractional (one fifth - 0.1mL) doses of IPV (fIPV) has become a very important focus. The approach is not new, having been assessed in trials undertaken in vaccine-naive infants, in OPV-primed infants and children, as well as in adults. In addition, given the practical and logistical challenges of needle and syringe (N&S)-based ID vaccine administration, the use of needle-free administration devices has also been explored previously.

In these trials, the administration of one fifth of a full dose by the ID route has consistently demonstrated a good safety profile. The rates of local reactions related to the administration of the vaccine by the ID route compared to the intramuscular (IM) route are higher in some although not in other trials. However, those reactions reported are generally mild and self-limiting irrespective of the method of administration employed. No significant systemic reactions or serious adverse events (SAE) related to ID fIPV administration have been reported. Furthermore, although when comparisons have been undertaken, the seroconversion rates and neutralizing antibody titres generated by the ID fIPV are consistently lower than those generated by a full IM dose of the same vaccine, the immunogenicity is such that the approach is viewed as a viable alternative in the context of the current Global Polio Eradication Initiative (GPEI) strategy.

Of particular importance, in studies undertaken in Cuba and Bangladesh, the administration of a single ID fIPV dose to poliovirus-vaccine naive infants has been shown to effectively prime the immune system for a subsequent rapid anamnestic response to an ID fIPV booster. In Cuba, priming with ID fIPV at four months of age resulted in a response within seven days of a subsequent ID fIPV booster dose at eight months - resulting in a cumulative seroconversion rate of 98% for poliovirus serotype 2 over the two dose course . The equivalent figure was 81% following a six and 14 week prime-boost schedule in Bangladesh. In both cases, the cumulative seroconversion rate following two ID fIPV doses was significantly higher for all serotypes than the seroconversion rate recorded following a single full-dose of IPV administered by the IM route (98% versus 62% in Cuba; 80% versus 39% in Bangladesh for serotype 2). The demonstrated anamnestic responses described, provide an effective strategy for rapidly inducing seroprotection in a primed population through the campaign-based provision of a second dose of ID fIPV - initiated as part of an OBR. In addition, if coverage can be assured, the use of a two dose ID fIPV routine schedule provides higher levels of seroprotection than a single IM IPV dose while still remaining dose sparing (0.2mL versus 0.5mL).

Based on the data available and their assessment of the current global landscape, the latest WHO position paper on polio vaccines, published in March 2016, suggests that '...countries could consider instituting a 2-dose fractional dose schedule, which could ensure that all eligible infants receive IPV...'. The same paper indicates that 'One fractional-dose IPV may be particularly appropriate for outbreak response if supplies are limited'. Based on this recommendation, and their own assessment, several states in India have subsequently decided to introduce two ID fIPV doses into their routine immunization schedule.

Rationale

While the safety and immunogenicity of ID fIPV is established in a clinic setting, there are little data examining the feasibility of rapid ID fIPV delivery in community-based campaign.

Many countries across sub-Saharan Africa, and other parts of the world where OPV supplementary immunization activities (SIA) are ongoing, have an established and highly effective framework for the campaign-based delivery of oral vaccines and other orally administered interventions (e.g. vitamin A and medendazole). However, such SIA commonly rely on the use of non-clinically trained individuals for frontline delivery (for example, volunteers from youth groups and other community organizations play a key role in such campaigns in The Gambia).

National campaigns involving the delivery of IM vaccines (e.g. MenAfriVac™ and most recently the measles and rubella combined vaccine [90-95% coverage of 802 425 target nine-month to 15 year olds in The Gambia in April 2016]) have also been undertaken very successfully - in this case relying on nurses and public health officers (or other health professionals involved in the routine provision Expanded Programme on Immunization (EPI) schedule) to administer the vaccines. However, the delivery of IM injections is part of the routine day-to-day practice of such professionals and can be completed with almost 100% success following limited training.

In contrast, the reliable delivery of ID injections, as is required to ensure the consistent immunogenicity of fIPV, is notoriously difficult with a N&S, particularly in active infants and children, and requires not only training but also significant practical experience. Indeed, data from both Cuba and The Gambia highlight that the immunogenicity of ID fIPV is directly determined by injection quality, as assessed by both ID bleb size and fluid loss at the injection site ([14] and The Gambia - unpublished data). Furthermore, given the nature of the injection, the approach is more time consuming than an IM vaccination (The Gambia - Figure 1 [unpublished data]) and markedly more time consuming than the delivery of a dose of OPV. This has important manpower implications even assuming personnel with the requisite skills are available.

Given these challenges, this pragmatic trial will specifically compare the feasibility of ID fIPV delivery using three different methods of administration in a campaign setting in rural part of The Gambia:

* Needle and syringe [N&S] (auto-disable, fixed needle)
* Intradermal Adapter [IDA] - West Pharmaceutical Services Inc
* Tropis™ Disposable Syringe Jet Injector [DSJI] - Pharmajet

Gaining an understanding of the utility of different methods of ID fIPV delivery in a campaign represents an important final step before key decisions regarding the approaches taken to fIPV delivery, particularly in an OBR, are finalized. A number of qualitative and quantitative endpoints will be assessed related to the practicalities of implementation. Information on solicited local and systemic reactogenicity will also be collected to strengthen the existing data set with this regard particularly related to campaign-based administration. Immunogenicity data will also be generated in a subset of 24 to 59 month old vaccine recipients to ensure that any factors enhancing the speed and ease of ID fIPV administration do not significantly compromise the ID fIPV immunogenicity - for example as a result of poor injection quality. This age group is chosen to limit the potential confounding effects of having received a different number of OPV and/or IPV doses present in younger age groups.

The data will also expand what is currently a very limited data-set regarding ID fIPV administration in sub-Saharan Africa - a setting where the risks of future cVDPV2 outbreaks is not inconsiderable despite recent sustained progress.

ELIGIBILITY:
Inclusion Criteria:

* Written or thumb-printed informed consent obtained from a child's parent or guardian
* Resident within the geographical area which is expected to be covered by the campaign
* Between 4 and 59 months of age at the time of the campaign

Exclusion Criteria:

* Anaphylaxis or a severe, potentially life threatening, allergic reaction to a previous vaccination
* Any other condition or significant acute illness meaning that it is judged to be against the infant's or child's best interests to receive ID fIPV (note that most chronic illnesses and minor acute illnesses - when normal vaccinations would be encouraged, do not represent exclusions for the trial)

Ages: 4 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2721 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
Total time taken to deliver ID fIPV using each of the three methods of administration | Collected on day 1, 2 or 3 of the vaccination campaign
Qualitative measures of administration method utility | Collected on day 1, 2 or 3 of the vaccination campaign
  Ergonomic characteristics of the intradermal administration methods collected through questionnaires
Local and systemic reactogenicity collected according to standard severity score (0 - 4) system. | Day 3 following vaccination
  Local reactogenicity (induration, erythema, tenderness, fever, vomiting, diarrhoea, feeding, irritability) will be collected on all vaccines on day 3 following vaccine administration
Serious adverse events (SAE) and adverse events (AE) following ID fIPV administration | Within 4 weeks of vaccination
Semi-quantitative measure of distress in infants and children associated with ID fIPV administration | Collected on day 1, 2 or 3 of the vaccination campaign
  Infant distress will be graded according to a visual analogue scale
Storage volumes of equipment required for ID fIPV delivery and subsequent bio-waste disposal including any differences the equipment required to safely deliver such vaccinations in a campaign | Collected on day 1, 2 or 3 of the vaccination campaign
  The volume of the disposables and biowaste created by each of the administration methods will be recorded.
Number of ID fIPV doses deliverable per IPV vial using each of the three administration methods (to identify any wastage associated with syringe/device filling) | Collected on day 1, 2 or 3 of the vaccination campaign
Immune response to ID fIPV (poliovirus neutralization assays) | Serum sample taken at baseline (pre-vaccination) and 4 weeks following vaccination
  Poliovirus neutralization assays
Changes in the time taken to deliver the ID fIPV and in the immune responses generated over the course of a 3 day campaign | Over 3 days of the campaign
Changes in the vaccine vial monitors (VVM) and also temperature deviations identified using a continuous temperature data logger associated with a campaign using each of the three administration methods | Over 3 days of the campaign
Qualitative factors which might influence campaign uptake in The Gambia and comparable sub-Saharan African settings | 1 week following vaccination campaign
Number of ID fIPV doses delivered using each of the three methods in the course of a defined campaign day by one vaccination team | Collected on day 1, 2 or 3 of the vaccination campaign

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MRCPCH MSc PhD, Principal Investigator — MRC Unit The Gambia; Adedapo O Bashorun, MBBS, Principal Investigator — MRC Unit The Gambia
Locations (1):
- MRC Unit The Gambia, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bashorun AO, Badjie Hydara M, Adigweme I, Umesi A, Danso B, Johnson N, Sambou NA, Fofana S, Kanu FJ, Jeyaseelan V, Verma H, Weldon WC, Oberste MS, Sutter RW, Jeffries D, Wathuo M, Mach O, Clarke E. Intradermal administration of fractional doses of the inactivated poliovirus vaccine in a campaign: a pragmatic, open-label, non-inferiority trial in The Gambia. Lancet Glob Health. 2022 Feb;10(2):e257-e268. doi: 10.1016/S2214-109X(21)00497-6. Epub 2021 Dec 21. PMID 34951974